CLINICAL TRIAL: NCT02316626
Title: Subcutaneous Progesterone Versus Vaginal Progesterone Gel for Luteal Phase Support in Gonadotropin Ovarian Stimulation for Intrauterine Insemination: a Pilot Randomized Controlled Study
Brief Title: Subcutaneous Progesterone Versus Vaginal Progesterone Gel for Luteal Phase Support
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Roberta Venturella (Other)
Responsible Party: Sponsor-Investigator, Roberta Venturella, MD, PhD Student, University Magna Graecia
Organization: University Magna Graecia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pleyris
Record Dates: First submitted 2014-12-07; First posted 2014-12-15 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subcutaneous progesterone (Experimental): Luteal phase support cycles will involve once-daily administration of 25 mg of SC P from the day after insemination for 14 days.
  Interventions: Drug: Subcutaneous progesterone
- Vaginal Progesterone (Active Comparator): Luteal phase support cycles will involve once-daily administration of 90 mg vaginal gel from the day after insemination for 14 days.
  Interventions: Drug: Vaginal progesterone

INTERVENTIONS:
Drug: Subcutaneous progesterone — 25 mg daily for 14 days
  Other Names: Pleyris
  Arms: Subcutaneous progesterone
Drug: Vaginal progesterone — 90 mg daily for 14 days
  Other Names: Crinone 8
  Arms: Vaginal Progesterone

SUMMARY:
It is well known that implantation of the developing blastocyst occurs during the luteal phase of the menstrual cycle when the endometrium is under the direct influence of Progesterone (P).Several prospective randomized controlled trials have evaluated the benefits of luteal phase P support in ovulation induction cycles and a recent review and meta-analysis demonstrated that it may be of benefit to patients undergoing ovulation induction with gonadotropins in intrauterine insemination (IUI) cycles. Until now, injectable P was offered only in an oil-base solution owing to the insoluble properties of the molecule, which made the IM route mandatory. A recent publication, however, demonstrated the efficacy of a new P formulation that could be a game changer. The aim of the present pilot trial will be to compare the efficacy and tolerability of 25 mg/d of the new SC P with 90 mg/d of vaginal gel P for luteal phase support (LPS) in COH and IUI cycles.

DETAILED DESCRIPTION:
The present randomized study will be conducted to compare the safety, effectiveness and tolerability of SC P (Pleyris; IBSA Institut Biochimique SA) with vaginal P gel (Crinone; Merck Serono) for LPS in COH/IUI cycles. The study will be conducted, recorded and reported in compliance with the principles of Good Clinical Practice (GCP) guidelines at the Department of Obstetrics and Gynecology of Magna Graecia University of Catanzaro.

ELIGIBILITY:
Inclusion Criteria:

<38 years of age with either primary or secondary infertility for at least 1 years; body mass index between 19 and 30 kg/m2; Day 2 serum FSH <15 IU/ml; normal serum prolactin level; normal uterine cavity on hysterosalpingography or hysteroscopy.-

Exclusion Criteria:

female partners with previous ovarian surgery, one ovary, polycystic ovaries on ultrasound examination, other endocrine abnormalities (i.e., polycystic ovarian syndrome, thyroid disorders, hyperprolactinemia, hypogonadotropic hypogonadism), diminished ovarian reserve (basal FSH level >15 IU/mL), or age of >38 years

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 246 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 8 weeks after IUI
  Number of patients with clinical pregnancy assessed by ultrasonography

SECONDARY OUTCOMES:
side effects | Women will be followed for the duration of treatment, an expected average of 14 days
  The side effects of Pleris (local reaction at the injection site) or Crinone treatment (vaginal irritation, inflammation, itching, leakage, and bleeding), as well as the systemic side effects (e.g., nausea, dizziness, breast pain) will be of particular interest and considered as secondary outcomes (tolerability).

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, MD,PhD, Study Director — Magna Graecia University of Catanzaro; Roberta Venturella, MD, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro, Catanzaro, Italy